CLINICAL TRIAL: NCT04448795
Title: Significance of Drain Amylase Levels After Pancreaticoduodenectomy
Brief Title: Impact of Highest Drain Fluid Amylase Levels on Surgical Outcomes and Postoperative Interventions in Patients Undergoing Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202000980B0
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Pancreas; Fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigated the impact of highest drain fluid amylase (DFA) level on postoperative pancreatic fistula (POPF) severity and outcomes of patients undergoing pancreaticoduodenectomy (PD) with POPF. Patient demographics of biochemical POPF and clinically relevant POPF (CR-POPF) were compared. Predictive factors were assessed using binary logistic regression. Receiver operating characteristic curve analysis was performed to determine the optimal cutoff value of highest DFA (beyond 3 days post-PD). The investigators compared length of hospital stay, surgical mortality rates, and need for postoperative interventions by highest DFA level.

ELIGIBILITY:
Inclusion Criteria:

* underwent PD from October 2010 to September 2018 in our institution

Exclusion Criteria:

* younger than 20 years of age
* clinical information was unavailable due to private or legal issues
* receiving PD without pancreaticojejunostomy

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: underwent PD in Chang Gung Memorial Hospital at Linkou
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
postoperative pancreatic fistula | through study completion, an average of 2 month
  fluid output of any measureable volume via an operatively placed drain with amylase activity greater than 3 times the upper normal serum value

SECONDARY OUTCOMES:
postoperative interventions | through study completion, an average of 2 month
  transarterial embolization, image-guided second drainage, and reoperation
length of hospital stay | through study completion, an average of 2 month
30-day mortality rates | 30 day

IPD SHARING:
Plan to Share IPD: No